CLINICAL TRIAL: NCT05062278
Title: Vinblastine Versus Oral Hydroxiurea in Newly Diagnosed AML With Hyperleukocytosis: a Phase 2 Clinical Study
Brief Title: Vinblastine for Leukoreduction in Newly Diagnosed AML and Hyperleukocytosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Head of Hematology Department, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE21-00019
Record Dates: First submitted 2021-07-26; First posted 2021-09-30 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: AML; Hyperleukocytosis
MeSH Terms: interventions — Vinblastine; Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnose AML will be allocated 1:1 to recieve single dose vinblastine or daily oral hydroxiurea
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous Vinblastine (Experimental): Single dose intravenous vinblastine (6mg/m2) in bolous.
  Interventions: Drug: Vinblastine
- Oral Hydroxiurea (Active Comparator): Patient will recieve oral hydroxiurea at a dose of 50mg/kg/day until response or administration of induction chemotherapy
  Interventions: Drug: Hydroxyurea capsules

INTERVENTIONS:
Drug: Vinblastine — Single-dose of intravenous vinblastine at 6mg/m2 (maximum 10mg).
  Other Names: Blestinib
  Arms: Intravenous Vinblastine
Drug: Hydroxyurea capsules — Oral hydroxyurea at a dose of 50mg/kg/day until the administration of induction chemotherapy.
  Arms: Oral Hydroxiurea

SUMMARY:
Vinblastine can leukoreduce patients with newly diagnosed AML and hyperleukocytosis but clinical trials are lacking.

DETAILED DESCRIPTION:
This phase 2 trial will explore the efficacy of a single dose of vinblastine (6mg/m2) to leukoreduce patients with newly diagnosed AML and hyperleukocytosis. Patients will be allocated 1:1 into two groups: intravenous single dose vinblastine or oral hydroxiurea (50mg/kg/day until response or induction chemotherapy). Effective leukoreduction and safety parameters will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Both genders
3. Diagnosis of non-M3 AML by the WHO 2016 diagnostic criteria
4. Patients eligible and not eligible for transplant
5. Patients eligible and not eligible for intensive treatment
6. AML secondary to treatment or associated to myelodisplasia
7. Leukocytes ≥50x106/L
8. Not being able to receive chemotherapy in the next two days

Exclusion Criteria:

1. AML with PMP/RAR-alfa translocation t(15;17)
2. Poor functional status (ECOG>2)
3. Active infection
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a significant reduction in the number of leukocytes by complete blood count | 2 days
  The proportion of patients with a reduction in the number of leukocytes higher than 50% by complete blood count at 48 hours after the intervention.

SECONDARY OUTCOMES:
Description of daily leukocytes by complete blood count after intervention | 5 days
  Document daily changes in the number of leukocytes by complete blood count after the administration of intravenous vinblastine or oral hydroxyurea.
Time to achieve a significant reduction in leukocyte count by complete blood count | 5 days
  Document time for effective leukoreduction by complete blood count after each intervention (defined as a reduction of >50% of leukocytes after intervention).

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Hopsital Universitario Dr. Jose E. Gonzalez, Centro Universitario contra el Cancer, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuo KH, Callum JL, Panzarella T, Jacks LM, Brandwein J, Crump M, Curtis JE, Gupta V, Lipton JH, Minden MD, Sher GD, Schimmer AD, Schuh AC, Yee KW, Keating A, Messner HA. A retrospective observational study of leucoreductive strategies to manage patients with acute myeloid leukaemia presenting with hyperleucocytosis. Br J Haematol. 2015 Feb;168(3):384-94. doi: 10.1111/bjh.13146. Epub 2014 Oct 10. PMID 25303497
- [Background] Marbello L, Ricci F, Nosari AM, Turrini M, Nador G, Nichelatti M, Tedeschi A, Vismara E, Morra E. Outcome of hyperleukocytic adult acute myeloid leukaemia: a single-center retrospective study and review of literature. Leuk Res. 2008 Aug;32(8):1221-7. doi: 10.1016/j.leukres.2008.01.004. Epub 2008 Mar 3. PMID 18313749
- [Background] Mamez AC, Raffoux E, Chevret S, Lemiale V, Boissel N, Canet E, Schlemmer B, Dombret H, Azoulay E, Lengline E. Pre-treatment with oral hydroxyurea prior to intensive chemotherapy improves early survival of patients with high hyperleukocytosis in acute myeloid leukemia. Leuk Lymphoma. 2016 Oct;57(10):2281-8. doi: 10.3109/10428194.2016.1142083. Epub 2016 Feb 5. PMID 26849624
- [Background] Salerni BL, Bates DJ, Albershardt TC, Lowrey CH, Eastman A. Vinblastine induces acute, cell cycle phase-independent apoptosis in some leukemias and lymphomas and can induce acute apoptosis in others when Mcl-1 is suppressed. Mol Cancer Ther. 2010 Apr;9(4):791-802. doi: 10.1158/1535-7163.MCT-10-0028. Epub 2010 Apr 6. PMID 20371726
- [Background] Sauter C, Fehr J, Frick P, Gmuer J, Honegger H, Martz G. Acute myelogenous leukemia: successful treatment of relapse with cytosine arabinoside, VP 16-213, vincristine and vinblastine (A-triple-V). Eur J Cancer Clin Oncol. 1982 Aug;18(8):733-7. doi: 10.1016/0277-5379(82)90071-2. PMID 6961036